CLINICAL TRIAL: NCT04053335
Title: Eliminating Low-Value Care in Virginia: Six Large Health Systems
Brief Title: Smarter Care Virginia, Examining Low-Value Care in Virginia
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, John N. Mafi, MD, MPH, Principal Investigator, University of California, Los Angeles
Other Study IDs: 75486025
Record Dates: First submitted 2019-08-05; First posted 2019-08-12 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Chronic Kidney Diseases; Eye Diseases; Cardiac Disease; Surgery; Low Back Pain
MeSH Terms: conditions — Renal Insufficiency, Chronic; Eye Diseases; Heart Diseases; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Multicomponent Physician Performance Peer-Comparison: Cohort 1 (6 groups):
  Inova/Signature Parters, Sentara/Sentara Quality Care Network, Ballad Health, Carilion Clinic, Health Care Associates Virginia/Virginia Care Partners, and Virginia and Commonwealth University Health System
  Note that the original design for the intervention was a step-wedge randomization. However, this was changed due to the COVID-19 pandemic, which necessitated a delay in all study activities from March 2020 - September 2020. The intervention began in September 2020. Data collection concluded in December 2022.
  Interventions: Behavioral: Multicomponent Physician Performance Peer-Comparison Feedback Intervention
- Cohort 2: Multicomponent Physician Performance Peer-Comparison: Cohort 2 (6 groups): Six comparable control health systems identified via matching

INTERVENTIONS:
Behavioral: Multicomponent Physician Performance Peer-Comparison Feedback Intervention — The intervention will consist of 5 components delivered simultaneously
  * Clinical Leadership Team: Each site will develop a Clinical Leadership Team (CLT), typically consisting of quality officers, clinician champions, etc. to implement and monitor the intervention
  * Speaker Series: VCHI will offer the CLTs access to national experts via a CME-approved speaker series and "office hours" to support the intervention.
  * Education Materials: The CLTs will distribute clinician and consumer education throughout the health systems calling to avoid 9 low-value services.
  * Clinician Report Cards: VCHI will distribute quarterly customized clinician performance report cards to the CLTs teams using the Milliman Health Waste Calculator and Virginia APCD
  * Quality improvement training: The intervention will provide the CLTs with in-person quality improvement and clinician performance feedback training, using principles of self-determination theory, and will include monthly check-in calls
  Groups: Cohort 1: Multicomponent Physician Performance Peer-Comparison

SUMMARY:
Low-value care is defined as patient care that provides no net benefit to patients in specific clinical scenarios, and can cause patient harm. Prior research has documented high-rates of low-value care in Virginia; this work has helped to inspire a Virginia government-sponsored quality improvement initiative to reduce low-value care. Funded by an Arnold Ventures grant, six large health systems in Virginia volunteered to partner with the Virginia Center for Health Innovation (VCHI) to reduce use of nine low-value health services (three preoperative testing measures, two cardiac screening measures, one diagnostic eye imaging measure, one low-back pain opioid measure, one low-back pain imaging measure and one peripherally inserted central catheter [PICC] measure). These health systems include nearly 7000 clinicians practicing across more than 1000 sites.

VCHI is implementing a nonrandomized physician peer-comparison feedback quality improvement intervention to reduce use of nine low-value services. Modeling will be used to identify and use propensity score matching to match six intervention health systems to six comparable control health systems. VCHI will provide education, quality improvement training and financial resources to each site, and VCHI will use the Milliman MedInsight Health Waste Calculator to create the peer comparison reports using the Virginia All Payer Claims Database (APCD). VCHI will use additional measures from The Agency for Healthcare Research and Quality (AHRQ). Additionally, VCHI will use AHRQ data to attribute physicians and health care facilities to health systems.

The primary purpose of the initiative is to improve quality of care for Virginia residents and this initiative is not being done for research purposes. Nevertheless, University of California, Los Angeles (UCLA) plans to rigorously study and publish the impact of this intervention across the state of Virginia, which is why the UCLA team pre-registered the initiative. The UCLA team will use the Virginia APCD to evaluate the impact of the intervention. Please note: the APCD has a 1-year time-lag of data collection and is a dynamic database, meaning that its population of enrollees changes from year to year. This intervention was initially designed as a randomized step-wedge intervention; the intervention was delayed by the COVID-19 pandemic and began in September 2020 for all intervention groups. The intervention period was extended through December 2022. As a result, the initial design was modified.

ELIGIBILITY:
Inclusion Criteria

All adult patients (aged 18 or older) at each of the six health systems who are at risk for receiving low-value care across each of the nine measures.

* For preoperative testing, eligible patients include those with a health system evaluation and management visits 30 days prior to low-risk surgery.
* For eye imaging, eligible patients will be patients with evaluation and management visits with a health system ophthalmologist/optometrist.
* For cardiac screening, eligible patients are patients with an ambulatory evaluation and management visit (all specialties).
* For the PICC line measure, eligible patients would include hospitalized patients.
* For the low-back pain measures, eligible patients include those who have a diagnosis of low-back pain or acute low-back pain.

Exclusion Criteria

* Patients under the age of 18.
* Patients who do not meet the above criteria.
* Patients who do not receive care at each of the six health systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients who receive care at six large health systems (and their three clinically integrated networks) in Virginia: (1) Ballad Health, (2) Carilion Clinic, (3) Hospital Corporation of America and Virginia Care Partners, (4) Inova and Signature Partners (Inova/Signature Patners will not be in main analysis) (5) Sentara Health System and Sentara Quality Care Network, (6) and Virginia Commonwealth University Health System.
Sampling Method: Non-Probability Sample
Enrollment: 5000000 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with low-value utilization across the 9 low-value care measures | 36 months
  Measures defined using evidence-based guidelines such as the USPSTF, American College of Cardiology, Choosing Wisely and others.
  The primary measure is global percentage of use among eligible patients across 9 measures (see eligibility criteria for measure-specific denominators):
  * Preoperative laboratory testing
  * Preoperative EKGs, chest x-rays and pulmonary function testing
  * Preoperative cardiac imaging/stress testing
  * Annual EKG/other cardiac screening for low-risk adults
  * Cardiac stress imaging/cardiac imaging in low-risk adults
  * Diagnostic eye imaging in low-risk patients
  * Peripherally inserted central catheters in stage 3-5 chronic kidney disease patients without nephrology consult
  * Opioid prescribing for low back pain (added Jan 2022)
  * Imaging for nonspecific low back pain (added Jan 2022)
  UCLA statisticians will independently assess measures using the Virginia APCD, which includes paid claims for Commercial, Medicaid, and Medicare insured patients

SECONDARY OUTCOMES:
Percentage participants with high-value utilization across the 9 measures (e.g., balancing measures) | 36 months
  These balancing measures will assess the use of high-value services. For example, the UCLA team will assess whether symptomatic (e.g., chest pain) patients continue to receive testing (e.g., EKGs) prior to low-risk surgery, or whether patients with eye disease continue to receive eye imaging, etc.
Percentage of participants with adverse events (e.g., peri-operative medical complications) | 36 months
  While VCHI, the UCLA team, and health systems do not expect adverse events (AEs) to increase in this evidenced-based quality improvement initiative, the UCLA team will monitor for them. AEs will be measure specific. For example, patients with preoperative visits will be evaluated for 30 day peri/post-operative medical complications (e.g., myocardial infarction). Patient eligible to receive cardiac screening (and do not receive it) will be evaluated for 30-day myocardial infarction diagnoses and hospitalization rates. Patients eligible to receive eye imaging and do not receive it will be evaluated for 1-year eye disease progression or new diagnosis rates. Patients eligible to receive a PICC line and do not will be evaluated for 30-day readmission rates. Each local health system QI team will also be provided education on how careful, nuanced attention to guidelines can reduce the risk of potential AEs.
Reduction in low- and high-value services by socioeconomic status | 36 months
  We will also assess for unintended consequences with an equity lens. For example, we will assess whether reductions in the high-value care measures disproportionately affected socioeconomically disadvantaged populations (e.g., those living in vulnerable neighborhoods or those with Medicaid insurance)
Total costs (estimates from percent effort of clinical leadership team, utilization trends | 36 months
  The cost analysis will estimate costs based on changes in utilization over time using costs as defined by the total amount paid to each provider (including out-of-pocket costs) available in the Virginia APCD. The UCLA team will also estimate the percent effort of each member of the clinical leadership team during the study time-frame to estimate investment costs. These latter data will be obtained via surveys and/or interviews of the clinical leadership teams.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No